CLINICAL TRIAL: NCT01081691
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CNTO 5825 Following a Single Intravenous or a Single Subcutaneous Administration in Healthy Subjects
Brief Title: A Study Evaluating Intravenous and Subcutaneous Administration of a Human Monoclonal Antibody (CNTO 5825) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sr. Director, CPTM, Centocor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015574; EudraCT No.: 2009-013343-11
Record Dates: First submitted 2010-02-18; First posted 2010-03-05 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: CNTO 5825; Safety; Phase I; Healthy adults; Healthy Atopic adults
MeSH Terms: interventions — CNTO 5825

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (7):
- 001 (Experimental): CNTO 5825 0.1 mg/kg single dose Intravenously (IV) or matching placebo
  Interventions: Biological: CNTO 5825
- 002 (Experimental): CNTO 5825 0.3 mg/kg single dose IV or matching placebo
  Interventions: Biological: CNTO 5825
- 003 (Experimental): CNTO 5825 1 mg/kg single dose IV or matching placebo
  Interventions: Biological: CNTO 5825
- 004 (Experimental): CNTO 5825 3 mg/kg single dose IV or matching placebo
  Interventions: Biological: CNTO 5825
- 005 (Experimental): CNTO 5825 10 mg/kg single dose IV or matching placebo
  Interventions: Biological: CNTO 5825
- 006 (Experimental): CNTO 5825 For atopic patient:10 mg/kg single IV dose or matching placebo
  Interventions: Biological: CNTO 5825
- 007 (Experimental): CNTO 5825 For atopic patient: 3 mg/kg single dose SC or matching placebo
  Interventions: Biological: CNTO 5825

INTERVENTIONS:
Biological: CNTO 5825 — 10 mg/kg single dose IV or matching placebo
  Arms: 005
Biological: CNTO 5825 — 3 mg/kg single dose IV or matching placebo
  Arms: 004
Biological: CNTO 5825 — For atopic patient:10 mg/kg single IV dose or matching placebo
  Arms: 006
Biological: CNTO 5825 — For atopic patient: 3 mg/kg single dose SC or matching placebo
  Arms: 007
Biological: CNTO 5825 — 0.3 mg/kg single dose IV or matching placebo
  Arms: 002
Biological: CNTO 5825 — 0.1 mg/kg single dose Intravenously (IV) or matching placebo
  Arms: 001
Biological: CNTO 5825 — 1 mg/kg single dose IV or matching placebo
  Arms: 003

SUMMARY:
The purpose of this study is to assess the safety and tolerability of CNTO 5825 following a single intravenous (IV) or subcutaneous (SC) dose administration in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), placebo controlled, double-blind (neither physician or subject knows the name of the assigned study medication) study to assess the safety, tolerability, immune response, pharmacokinetics (what the body does to the drug), and pharmacodynamics (what the drug does to the body) of CNTO 5825. The study population will consist of 48 healthy volunteers and 16 healthy atopic volunteers. Five dose levels of study agent will be assessed. Participants will be required to stay at the research center after study agent administration for the inpatient portion of the study and then return for out-patient visits. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events. Placebo (containing inactive substances only) or one of five dose levels of CNTO 5825 will be given. Healthy volunteers will be given a single IV infusion (directly into a vein) or a single dose of up to 3 injections under the skin. Healthy atopic volunteers will be given one dose as as an IV infusion. There will be a screening period of up to 4 weeks. All participants will be in the study for 17 weeks after dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman with no clinically significant abnormalities
* Body weight in the range of 50 to 100 kg inclusive
* Body mass index (BMI) of 18.5 to 30 kg/m2 inclusive
* For healthy atopic patients: history of atopic allergy

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to any biologic medication or to any components of the formulation used in this study
* Received an experimental antibody or biologic therapy within the previous 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CNTO 5825 by evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events in healthy volunteers. | 17 weeks post dose

SECONDARY OUTCOMES:
Evaluate the effects of CNTO5825 on the body and the effects of the body on CNTO 5825 (Pharmacokinetics (PK), Pharmacodynamics (PD)) | 17 weeks post dose
Immune response (Immunogenicity) after dose with CNTO 5825 | 17 weeks post dose

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Derived] van Hartingsveldt B, Nnane IP, Bouman-Thio E, Loza MJ, Piantone A, Davis HM, Petty KJ. Safety, tolerability and pharmacokinetics of a human anti-interleukin-13 monoclonal antibody (CNTO 5825) in an ascending single-dose first-in-human study. Br J Clin Pharmacol. 2013 May;75(5):1289-98. doi: 10.1111/j.1365-2125.2012.04477.x. PMID 23043368